CLINICAL TRIAL: NCT06516471
Title: The Evolution of Safety and Efficacy of Neuroendoscopy Guided by Head-mounted Mixed Reality Technique Navigation System for Tumor Resection in Pineal Region and Brainstem: A Prospective, Randomized, Parallel-controlled Clinical Study
Brief Title: The Evolution of Neuroendoscopy Guided by Head-mounted Mixed Reality Technique Navigation System in Neurosurgery
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: B2024-192
Record Dates: First submitted 2024-06-21; First posted 2024-07-24 (Actual); Last update posted 2024-07-24 (Actual); Status verified 2024-07

CONDITIONS: Pineal Tumor; Brainstem Tumor; Surgery
MeSH Terms: conditions — Pinealoma; Brain Stem Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mixed Reality Navigation System Group (Experimental): Patients will receive receive surgery guided by mixed reality technique navigation system.
  Interventions: Device: Conventinal Navigation System Group
- Conventinal Navigation System Group (Active Comparator): Patients will receive receive surgery guided by traditional navigation system.
  Interventions: Device: Conventinal Navigation System Group

INTERVENTIONS:
Device: Conventinal Navigation System Group — The preoperative planned model is projected onto the endoscopic display area in 3D using a mixed reality headset, accurately matching the actual anatomical structure and tissue displayed under the patient's endoscope to guide surgical resection of tumors.

SUMMARY:
The pineal region and brainstem tumors are located at the central position of the cranial cavity, surrounded by important neural structures and venous systems, leading to challenges in preoperative diagnosis, adding uncertainty and complexity to treatment. For a long time, surgical treatment of pineal region and brainstem tumors has been one of the most challenging areas in neurosurgery.

With the development of neuroendoscopy and virtual endoscopy technologies, how to convert complex three-dimensional bone, vascular, and neural images into virtual endoscopic images and how to combine virtual endoscopy with neuro-navigation for endoscopic skull base surgery to provide high-quality guidance images for surgery has become an urgent new research issue.

The project team plans to develop a neuroendoscopy combined with a wearable mixed reality glasses navigation system, integrating the advantages of wearable glasses and existing surgical navigation systems.

This study aims to evaluate the role of mixed reality navigation systems in improving total resection and reducing major complications in patients with pineal region and brainstem tumors, as well as shortening surgical times.

DETAILED DESCRIPTION:
The pineal region and brainstem tumors are located at the central position of the cranial cavity, surrounded by important neural structures and venous systems. They contain many crucial neural functional nuclei, making surgical exposure and resection difficult. Furthermore, the tumors in this region exhibit complex and diverse pathological types, including mixed tumors, leading to challenges in preoperative diagnosis, adding uncertainty and complexity to treatment. Pineal region tumors commonly cause obstructive hydrocephalus, resulting in severe preoperative intracranial hypertension symptoms, further complicating surgical management. For a long time, surgical treatment of pineal region and brainstem tumors has been one of the most challenging areas in neurosurgery.

With the development of neuroendoscopy and virtual endoscopy technologies, how to convert complex three-dimensional bone, vascular, and neural images into virtual endoscopic images and how to combine virtual endoscopy with neuro-navigation for endoscopic skull base surgery to provide high-quality guidance images for surgery has become an urgent new research issue.

The project team plans to develop a neuroendoscopy combined with a wearable mixed reality glasses navigation system, integrating the advantages of wearable glasses and existing surgical navigation systems. While ensuring the accuracy of the navigation system, the team aims to fundamentally change the output method of the system, enabling the surgical navigation system to go beyond mere validation of effects and truly play a role of "intuitive visual navigation." By holographically observing and tracking the relevant blood vessels and nerves in the patient's area, the team has achieved high-precision integration of virtual and real microanatomy structures, allowing for better and safer handling of deep-seated tumors under the endoscope. This study aims to evaluate the role of mixed reality navigation systems in improving total resection and reducing major complications in patients with pineal region and brainstem tumors, as well as shortening surgical times.

ELIGIBILITY:
Inclusion Criteria:

1. Preoperative suspicion of pineal region and brainstem tumors;
2. Age range from 18 to 70 years old;
3. Preoperative neurological function was good, with KPS>70 points;
4. Informed consent of patients and their families;

Exclusion Criteria:

1. Recurrent pineal region and brainstem tumors, previously received radiation therapy;
2. Combined with serious cardiovascular disease, other systemic malignancies, and other diseases;
3. Participants who participate in clinical trials of other drugs or devices but fail to achieve the main research endpoint;
4. The subjects are unable or unwilling to participate in this experiment
5. Preoperative discussion considers that patients are unable to undergo neurosurgical endoscopic surgery and require the use of microscopy or other techniques to assist in tumor resection;

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-07 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Surgical time | immedately after surgery
  From openning the dura mater to close it

SECONDARY OUTCOMES:
Gross total resection rate | within 72 hours after surgery
  Gross total was defined as 100% of tumor resection
The incidence of complications | within 1 month after surgery
  new cranial nerve dysfunction, secondary surgery

IPD SHARING:
Plan to Share IPD: Yes
Study protocol ，CRF
Supporting Information: Study Protocol, SAP, CSR
Time Frame: When final results reported